CLINICAL TRIAL: NCT04496076
Title: Severe Neurologic Injury Outcomes During COVID-19 Crisis
Brief Title: COVID-19 Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sherry Hsiang-Yi Chou, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY20030201
Record Dates: First submitted 2020-07-13; First posted 2020-08-03 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-04

CONDITIONS: Sars-CoV2; Severe Neurologic Injury; Ischemic Stroke; Hemorrhagic Stroke; Intracerebral Hemorrhage; Subarachnoid Hemorrhage; Traumatic Brain Injury; Status Epilepticus
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Cerebral Hemorrhage; Subarachnoid Hemorrhage; Brain Injuries, Traumatic; Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective cohort minimal risk study to determine the impact of the COVID-19 crisis on outcomes of neurologically injured ICU patients.

DETAILED DESCRIPTION:
COVID 19 pandemic has overwhelmed healthcare capacity in many regions around the world. As resources become more limited and we have to triage /ration ventilators, neurologically injured ICU patients without COVID 19 but with respiratory insufficiency may be triaged to no ventilator care due to their perceived or actual prognosis. This may lead to increased rates of withdrawal of care and mortality. Some neurologically injured ICU patients with respiratory insufficiency may be simultaneously infected with COVID 19. Their outcomes are completely unknown. Capturing data on the prevalence of limitation of care and prognosis in this patient population will provide important information towards ongoing efforts in patient care and resource utilization as we face the rapidly evolving COVID 19 pandemic. Given the expected strain on ICU resources and limitations in research in ICUs during COVID 19 pandemic, data capture/study design must be targeted and pragmatic. This study is designed to answer the most basic and important questions while minimizing the burden of data collection on already overloaded providers.

This study design is comprised of two components: Component 1- Prospective cohort prevalence study captures data related to treatments offered, limitations of care and patient outcome in 5 select primary neurological diagnoses requiring ICU care. Component 2- Case control study captures the same data elements in the same patient populations during the 3 months prior COVID 19 pandemic (Sept - Dec, 2019).

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 18
* Patients who require critical care with primary diagnoses of: Acute ischemic stroke (AIS), acute intracerebral hemorrhage (ICH), acute subarachnoid hemorrhage (SAH), acute traumatic brain injury (TBI), status epilepticus (SE) patients requiring critical care

Exclusion Criteria:

* Patients under the age of 18 years old
* Pre-existing Do Not Resuscitate (DNR), Do Not Intubate (DNI), or Comfort Measures Only (CMO) status prior to acute hospitalization
* Neurologically morbid-bound on hospital arrival (bilateral fix/dilated pupils, catastrophic bleed/TBI) and likely to progress to brain death within 48 hrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 5 select primary neurological diagnoses (Acute Ischemic Stroke, Acute Intracerebral Hemorrhage, Acute Subarachnoid Hemorrhage, Acute Traumatic Brain Injury, Status Epilepticus) requiring ICU care
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
In-hospital Mortality | At hospital discharge, approximately 1 month
30-day mortality | 30 days post-hospital discharge

SECONDARY OUTCOMES:
Limitations of patient care- Frequency of care not being provided | During In-hospital course, up to 1 month
  Care treatment such as ventilator use, intubation, and/or tracheostomy
Limitations of patient care- Conversion of DNR/DNI/CMO status | During In-hospital course, up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sherry H Chou, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No